CLINICAL TRIAL: NCT07360184
Title: The Effect of Laughter Yoga on Fear of Childbirth and Self-Efficacy During Childbirth in Primiparous Women: A Randomized Controlled Trial
Brief Title: The Effect of Laughter Yoga on Primiparous Pregnant Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Betül Bal, Lecturer Doctor, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ASYO
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Laughter
MeSH Terms: conditions — Laughter | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter (Experimental): group performing laughter yoga
  Interventions: Behavioral: Laughter yoga
- Control (No Intervention): group not receiving intervention

INTERVENTIONS:
Behavioral: Laughter yoga — Sessions will consist of warm-up and breathing exercises, guided intentional laughter exercises, diaphragmatic breathing and relaxation, followed by a short mindfulness and closing phase.
  Arms: Laughter

SUMMARY:
Primiparous women constitute a special risk group who may experience higher levels of fear of childbirth and lower birth self-efficacy during pregnancy due to their lack of prior childbirth experience. Fear of childbirth is associated with increased anxiety, negative birth experiences, and unnecessary medical interventions, while birth self-efficacy is an important determinant of adaptation to the birth process and positive birth outcomes. In recent years, non-pharmacological and mind-body-based interventions have become increasingly important in the management of these psychological problems. Laughter yoga is a complementary method that combines conscious laughter exercises with breathing techniques to reduce stress and anxiety. This randomized controlled trial aims to evaluate the effect of laughter yoga on fear of childbirth and self-efficacy during childbirth in primiparous pregnant women. The study aims to provide scientific evidence for the use of laughter yoga as an effective, safe, and inexpensive psychosocial intervention that can be applied in prenatal care.

DETAILED DESCRIPTION:
Primiparous pregnant women are considered a special risk group during pregnancy from a physical, psychological, and social perspective because they have not previously experienced childbirth. Primiparous pregnancy refers to a woman's first pregnancy, and during this process, women may experience more stress and psychological difficulties than multiparous women due to their lack of experience with childbirth, uncertainty, perceived loss of control, and concerns about the future. The literature indicates that primiparous women report higher levels of anxiety, stress, and psychological sensitivity during pregnancy, and that lack of knowledge and uncertainty about the birth process exacerbate these problems. For this reason, primiparous women are considered a priority group in terms of psychological support and protective interventions during the prenatal period.

One of the most commonly reported psychological problems in primiparous women is fear of childbirth. Fear of childbirth, defined in medical literature as tokophobia, is an intense fear of pregnancy and the birth process that can impair functioning and lead to avoidance behaviors. Studies show that primiparous pregnant women have significantly higher levels of fear of childbirth compared to multiparous women. This fear is related to expectations of labor pain, loss of control during childbirth, anxiety about medical interventions, and fears about possible complications. High levels of fear of childbirth can lead to negative outcomes in primiparous women, such as increased anxiety, prolonged labor, decreased satisfaction with childbirth, and increased requests for elective cesarean delivery without medical necessity. Furthermore, it has been reported that fear of childbirth can negatively affect mental health, mother-infant bonding, and breastfeeding in the postpartum period.

Another important concept closely related to fear of childbirth in primiparous women is self-efficacy in childbirth. Self-efficacy in childbirth refers to a woman's perceived confidence in her ability to cope with the physical and emotional challenges she will encounter during the birth process and is based on Bandura's self-efficacy theory. The literature shows that birth self-efficacy is lower in primiparous women than in multiparous women and that low self-efficacy levels are one of the key factors that increase fear of childbirth [6,11]. Primiparous women with low birth self-efficacy tend to believe that they will not be able to cope with labor pains, experience fear of losing control during birth, and develop negative expectations about childbirth. A study conducted in Turkey shows a significant and inverse relationship between perceived birth self-efficacy and fear of childbirth; it reveals that as self-efficacy increases, fear of childbirth decreases. These findings indicate that strengthening birth self-efficacy in primiparous women is an important goal in reducing fear of childbirth.

While pharmacological and medical approaches exist for managing fear of childbirth and low birth self-efficacy, non-pharmacological and complementary methods have gained increasing importance in recent years. One such method, laughter yoga, is a mind-body-based practice that combines conscious laughter exercises with breathing techniques. Laughter yoga is based on the principle that the brain does not distinguish between spontaneous and conscious laughter; it has been reported that even simulated laughter reduces stress hormones and increases endorphin release. The literature shows that laughter yoga has positive effects on stress, anxiety, and psychological well-being; it increases oxygenation, reduces muscle tension, and strengthens individuals' emotional resilience. In line with these mechanisms, laughter yoga is thought to reduce fear of childbirth in primiparous women, creating a more positive emotional state and strengthening the woman's self-confidence and birth self-efficacy.

The current literature includes studies examining the effects of yoga, relaxation exercises, and similar mind-body interventions during pregnancy on fear of childbirth and childbirth self-efficacy. There are also a limited number of randomized controlled trials showing the positive effects of laughter yoga on mental health, stress levels, and prenatal bonding during pregnancy. However, a review of the literature reveals no randomized controlled trials directly examining the effects of laughter yoga on fear of childbirth and self-efficacy during childbirth in primiparous pregnant women. This situation clearly demonstrates the need for studies that reveal the relationship between these variables and the potential effects of laughter yoga. This study aims to fill this important gap in the literature by evaluating the effects of laughter yoga on fear of childbirth and self-efficacy during childbirth in primiparous pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* never having given birth before
* be a primiparous pregnant woman experiencing her first birth,
* be pregnant with a single baby,
* be approximately 28-34 weeks pregnant at the start of the intervention,
* be planning a vaginal birth,
* have the ability to read and speak Turkish,
* volunteer to participate in the study

Exclusion Criteria:

* A diagnosis of high-risk pregnancy or the presence of serious obstetric complications that prevent participation in exercise (e.g., placenta previa, uncontrolled gestational hypertension or preeclampsia, bed rest recommended due to threatened preterm labor, cervical insufficiency),
* multiple pregnancy,
* history of recurrent pregnancy loss (≥2 miscarriages) or pregnancy achieved through assisted reproductive techniques (e.g., IVF),
* diagnosis of a known psychiatric disorder (major depression, anxiety disorder, psychosis, etc.),
* history of alcohol or substance use during pregnancy,
* Severe orthopedic problems or chronic respiratory system diseases that prevent participation in light exercise or laughter exercises,
* Participation in other structured prenatal interventions (e.g., prenatal yoga, hypno-birth, intensive childbirth education programs) aimed at reducing fear or anxiety about childbirth during the study period.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-22 (Estimated)

PRIMARY OUTCOMES:
Wijma Childbirth Expectation/Experience Questionnaire - Version A (W-DEQ/ Version A) | Baseline (Day 0) and Week 4
  It was developed by Klaas and Barbro Wijma to measure women's fear of childbirth. The scale consists of 33 items. Responses on the scale are numbered from 0 to 5 and are on a six-point Likert scale. 0 means "completely," and 5 means "not at all." The minimum score on the scale is 0, while the maximum score is 165. As the score increases, so does the fear of childbirth experienced by women. While the first version of the scale did not specify a score range, subsequent studies determined a scoring range. This range can be used when interpreting scale scores. The total item score is interpreted as 0-60 for low fear of childbirth, 61-84 for moderate fear of childbirth, and 85 and above for high fear of childbirth.

SECONDARY OUTCOMES:
Self-Efficacy Scale in Childbirth (SEB-C32) | Baseline (Day 0) and Week 4
  The Self-Efficacy Scale for Childbirth was developed by Lowe (1993) to assess women's confidence and coping ability during childbirth. The short version of the scale was later developed by Ip et al. The Turkish validity and reliability study was conducted by Ersoy, with a Cronbach's alpha coefficient of 0.90. The scale consists of two subscales-outcome expectation and efficacy expectation-each comprising 16 items. Total scores range from 32 to 320, with higher scores indicating greater self-efficacy for childbirth. Items are rated on a 10-point Likert scale, with higher scores reflecting higher perceived competence and positive outcome expectations.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdağmadeni School of Health, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No